CLINICAL TRIAL: NCT06735482
Title: Effect of Therapeutic Play Activities on Motor Adaptive Behavior in Egyptian Children With Mild Intellectual Disability
Brief Title: Therapeutic Play in Children With Mild Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tayseer Saber Abdeldayem, Dr, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPTBSUREC/0903/241124
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Intellectual Disability; Intellectual Disability, Mild; Motor and Developmental Delay; Motor Delay; Adaptive Behavior; Physical Disability
Keywords: Play; Play therapy; Therapeutic play; Motor Adaptive Behavior; Adaptive Behavior; Intellectual Disability
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular; Learning Disabilities; Psychomotor Disorders

STUDY DESIGN:
Intervention Model Description: Quasi experimental
Who Masked: Outcomes Assessor
Masking Description: The assessor is blinded for the assessed children's allocation in groups. in both preprogram and postprogram assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Experimental (Experimental): Therapeutic Play Activities program for children with mild intellectual disability.
  a program of therapeutic play activities aimed at improving the adaptive motor skills of children with intellectual disabilities. The program consists of 24 sessions of play-based activities that will be applied in 2 months on a day-by-day basis. Therapeutic Play programs include activities that address core strength, bilateral coordination, motor skills, visual skills, body awareness, outdoor sensory activities, vestibular, and balance skills. Activities will be simulated for the child by the therapist to ensure the child understands them.
  Interventions: Behavioral: Therapeutic play program
- Group B control (No Intervention): Children will not receive any intervention

INTERVENTIONS:
Behavioral: Therapeutic play program — Therapeutic Play programs include activities that address core strength, bilateral coordination, motor skills, visual skills, body awareness, outdoor sensory activities, vestibular, and balance skills.
  Other Names: play therapy program
  Arms: Group A Experimental

SUMMARY:
The aim of this study is to determine the effectiveness of a designed therapeutic play activities program on improving motor adaptive behavior in a sample of Egyptian children with mild intellectual disabilities. The main question it aims to answer is:

What is the effect of therapeutic play activities in improving adaptive motor skills (fine-gap) of children with mild intellectual disability? A quasi-experimental design will be used as researchers will compare therapeutic play exercise program to standard treatment to find its effect on motor adaptive behavior in the selected sample of children with mild intellectual disability

Participants will:

Take play-based activity program for 24 sessions in 2 months Have a pre- and post-intervention evaluation of motor adaptive behavior by Vineleand Adaptive Behavior Scale II

DETAILED DESCRIPTION:
The research sample consists of twenty children whose ages range between 5 and 9 years of children with mild intellectual disabilities, with intelligence coefficients ranging between 50 and 70 on the Stanford Binet Scale, 5th edition (SB-5). The sample will be divided into two groups: 10 children in the control group and 10 children in the experimental group.

Methods For Intervention Experimental group Therapeutic Play Activities program for children with mild intellectual disability The validation of the current research hypotheses required the preparation and design of a program of therapeutic play activities aimed at improving the adaptive motor skills of children with intellectual disabilities. The program consists of 24 sessions of play-based activities that will be applied in 2 months on a day-by-day basis. Therapeutic Play programs include activities that address core strength, bilateral coordination, motor skills, visual skills, body awareness, outdoor sensory activities, vestibular, and balance skills. Activities will be simulated for the child by the therapist to ensure the child understands them. All children will be evaluated by VABSII before and after implementation of the program.

ELIGIBILITY:
Inclusion Criteria:

The child should be between 5 and 9 years of age of both sexes

- The child should be of mild intellectual disabilities according to Stanford Binet scale 5th edition The child should not be suffering from any apparent physical deformity in upper limbs, lower limbs or spine The child should not suffer from any visual or auditory disorder

Exclusion Criteria:

Children out of age range Children with moderate or severe intellectual disabilities Children with physical deformities in upper limb, lower limb or spine Children suffering from visual or auditory disorders

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
The Stanford-Binet Scale, the fifth edition (SB-5) | 8 weeks
  The Stanford-Binet Scale, the fifth edition, aims to measure intelligence and cognitive abilities in humans, in the age range of (2-85 years).
The Vineland Adaptive Behavior Scale: Second Edition (Vineland II) | 8 weeks
  The Vineland Adaptive Behavior Scale II measures an individual's development of personal independence and social responsibility by gathering information about day-to-day activities necessary to take care of oneself and to get along with others.

CONTACTS AND LOCATIONS:
Overall Officials: Tayseer S Abdeldayem, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No